CLINICAL TRIAL: NCT01400932
Title: Study STF115288, a Clinical Confirmation Study of GI148512 (Benzoyl Peroxide 3% Gel) in the Treatment of Acne Vulgaris in Japanese Subjects.- A Multicenter, Randomized, Double-blinded, Vehicle-controlled, Parallel-group Study -
Brief Title: Study STF115288, a Clinical Confirmation Study of GI148512 in the Treatment of Acne Vulgaris in Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115288
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2012-05

CONDITIONS: Acne Vulgaris
Keywords: inflammatory lesion; Benzoyl peroxide (BPO); once daily; acne vulgaris; vehicle gel; clindamycin (CLDM) 1%-BPO 3% gel; non-inflammatory lesion
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GI148512 (Benzoyl Peroxide 3% Gel) (Experimental): Subjects will apply in a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin). Also, the dose regimen will be once daily in the evening/bedtime. Comparison of 2 arms (GI148512 vs vehicle)
  Interventions: Drug: GI148512
- vehicle gel (Placebo Comparator): Subjects will apply in a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin). Also, the dose regimen will be once daily in the evening/bedtime.
  Interventions: Drug: vehicle gel

INTERVENTIONS:
Drug: GI148512 — GI148512, Topical gel in 1 g containing benzoyl peroxide 30 mg
  Other Names: Benzoyl Peroxide 3% Gel
  Arms: GI148512 (Benzoyl Peroxide 3% Gel)
Drug: vehicle gel — Matching vehicle gel of GI148512, not containing active ingredient (benzoyl peroxide)
  Arms: vehicle gel

SUMMARY:
This is a multicenter, randomized, double-blinded, vehicle-controlled, parallel-group study in Japanese subjects with acne vulgaris to demonstrate the efficacy of GI148512 (benzoyl peroxide [BPO] 3% gel) when applied once daily for 12 weeks. This study will also evaluate the safety of GI148512 when applied topically once daily for 12 weeks.

DETAILED DESCRIPTION:
Main inclusion criteria will be 12 to 45 years of age, who have an Investigator Static Global Assessment (ISGA) score of 2 or greater at baseline visit, and have both 17 to 60 facial inflammatory lesions (papules plus pustules) and 20 to 150 facial non-inflammatory lesions (open and closed comedones), including nasal lesions. The primary objective is to demonstrate the superiority of GI148512 to vehicle gel in total lesion counts. The secondary objectives are to demonstrate the superiority of GI148512 to vehicle gel in inflammatory lesion counts, and to evaluate the efficacy of GI148512 compared with vehicle gel at each visit. A total of 360 subjects will be enrolled and randomly assigned to one of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 12 to 45 years (inclusive) of age in good general health.
* Subjects must have both on the face:

A) A minimum of 17 but not more than 60 inflammatory lesions (papules / pustules), including nasal lesions.

And B) A minimum of 20 but not more than 150 non-inflammatory lesions (open / closed comedones), including nasal lesions.

* An ISGA (global assessment of severity by the investigator: refer to Section 6.2.1 "Assessment") score of 2 or greater at baseline.
* Females of childbearing potential and women who are less than 2 years from their last menses must agree to use the contraception.
* The ability and willingness to follow all study procedures and attend all scheduled visits.
* The ability to understand and sign a written informed consent form (Written informed consent must be obtained also from the parent or guardian in case of subject under 20 years of age at the time of given consent).

Exclusion Criteria:

* Have any nodule-cystic lesions at baseline.
* Are pregnant or breast-feeding.
* Used any of the following agents on the face within the previous 2 weeks: Topical antibiotics (or systemic antibiotics); Topical anti-acne medications (e.g., BPO, azelaic acid, resorcinol, salicylates); Abradants, facials, or peels containing glycolic or other acids; Masks, washes or soaps containing BPO, sulfacetamide sodium, or salicylic acid; Non-mild facial cleansers (e.g., facial scrub, cleansers containing agents with anti-inflammatory action); Moisturizers that contain retinol, salicylic acid, or α- or β-hydroxy acids; Astringents and toner (Subjects are allowed to enroll in this study, if the subject has been on treatment for more than 2 consecutive weeks prior to start of investigational product use).
* Used the following agents on the face or performed the following procedure within the previous 4 weeks: Topical corticosteroids (Use of inhaled, intra-articular, or intra-lesional steroids other than for facial acne is acceptable); Facial procedure (such as chemical or laser peel, microdermabrasion, blue light treatment, etc.).
* Used systemic retinoids within the previous 6 months or topical retinoids on the face within the previous 6 weeks.
* Received treatment with estrogens, androgens, or anti-androgenic agents within the previous 12 weeks (Subjects who have been treated with the above agents for more than 12 consecutive weeks prior to start of investigational product are allowed to enrol as long as they do not expect to change dose, drug, or discontinue use during the study).
* Used any medication that in the opinion of the investigator may affect this clinical study or evaluation of the study.
* Plan to use medications that are reported to exacerbate acne (e.g., mega-doses of certain vitamins, such as vitamin D [>2000 IU/day] and vitamin B12 [>1 mg/day], corticosteroids*, androgens, haloperidol, halogens [e.g., iodide and bromide], lithium, hydantoin, and phenobarbital).

  *: except the using of topical corticosteroids (e.g., inhaled, intra-articular, or intralesional steroids) other than for facial acne.
* Have a known hypersensitivity or have had previous allergic reaction to any of the components of the investigational product.
* Used any investigational therapy within the previous 12 weeks, or plan to participate in another clinical study at the same time.
* Participated in Japanese clinical studies planned by GlaxoSmithKline K.K. in the development of investigational products for acne vulgaris.
* Are currently abusing drugs or alcohol.
* Have a significant medical history of being immunocompromised.
* People as follows and the family members; Employees of GlaxoSmithKline, contract research organization (CRO) or site management organization (SMO); Investigators.
* Have other conditions that would put the subject at unacceptable risk for participation in the study.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (4):
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- GI148512: Participants applied 2 finger tip units (FTU) of GI148512 topically once daily in the evening/bedtime, over the entire face (including the forehead, nose, cheeks, and chin), for a treatment period of 12 weeks.
- Vehicle Gel: Participants applied 2 FTU of matching vehicle gel of GI148512 without the active ingredient topically once daily in the evening/bedtime, over the entire face (including the forehead, nose, cheeks, and chin), for a treatment period of 12 weeks.
Period: Overall Study
Arm/Group | GI148512 | Vehicle Gel
Started | 178 | 182
Completed | 164 | 167
Not Completed | 14 | 15
Not completed — Adverse Event | 10 | 5
Not completed — Lack of Efficacy | 0 | 3
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Deviation | 0 | 1
Not completed — Met Protocol-defined Stopping Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GI148512: Participants applied 2 FTU of GI148512 topically once daily in the evening/bedtime, over the entire face (including the forehead, nose, cheeks, and chin), for a treatment period of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | GI148512 | Vehicle Gel | Total
Number analyzed (Participants) | 178 | 182 | 360
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.3 (5.93) | 22.4 (6.76) | 21.9 (6.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 116 | 234
  Male | 60 | 66 | 126
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian-Japanese Heritage | 178 | 182 | 360
Total Lesion Counts at Baseline [Mean (Standard Deviation); unit: lesion counts] — The investigator (or subinvestigator) counted all inflammatory lesions (papules, pustules, and nodular lesions) and non-inflammatory lesions (open and closed comedos; diagnosis based on palpation) on the face at each study visit.
  lesion counts | 72.1 (33.40) | 70.3 (30.89) | 71.2 (32.12)
Non-inflammatory Lesion (NIL) Counts at Baseline [Mean (Standard Deviation); unit: lesion counts] — The investigator/subinvestigator counted all non-inflammatory lesions (open and closed comedo) on the face at each study visit. An open comedo is an open, widely dilated follicle with black-colored sebum, due to melanin and oxidation, and keratinous material that forms a plug, thereby obstructing the pilosebaceous duct. A closed comedo is a closed follicle filled with impacted sebum covered by keratin that has a whitish color.
  lesion counts | 44.2 (28.03) | 42.7 (26.28) | 43.4 (27.14)
Inflammatory Lesion (IL) Counts at Baseline [Mean (Standard Deviation); unit: lesion counts] — The investigator/subinvestigator counted all inflammatory lesions (papules, pustules, and nodular lesions [NL]) on the face at each study visit. A papule is a small, raised, red, dome-shaped palpable lesion. A pustule is a raised, dome-shaped palpable lesion containing yellow fluid (pus). A nodule may be a raised or deep-seated, dome-shaped palpable lesion of at least 5 millimeters in diameter.
  lesion counts | 28.0 (10.76) | 27.5 (10.09) | 27.7 (10.41)
Participants with the Indicated Investigational's Static Global Assessment (ISGA) Score at Baseline [Number; unit: participants] — Investigators evaluated the acne severity of the participants' face using the ISGA scale, ranging from 0 to 5: 0=clear skin with no ILs or NILs; 1=almost clear: rare NILs with no more than rare papules; 2=mild acne: greater than Grade 1, some NILs with no more than a few ILs (papules/pustules only, no NLs); 3=moderate acne: greater than Grade 2, up to many NILs and had some ILs, but no more than one small NL; 4=severe acne: greater than Grade 3, up to many NILs and ILs, but no more than a few NLs; 5=very severe acne: many NILs and ILs and more than a few NLs, had cystic lesions.
  participants
    0: Clear | 0 | 0 | 0
    1: Almost Clear | 0 | 0 | 0
    2: Mild Severity | 41 | 45 | 86
    3: Moderate Severity | 117 | 118 | 235
    4: Severe | 20 | 19 | 39
    5: Very Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Total Lesion Counts From Baseline to Week 12
Description: The investigator (or subinvestigator) counted all inflammatory lesions (papules, pustules, and nodular lesions) and non-inflammatory lesions (open and closed comedos; diagnosis based on palpation) on the face at each study visit. An open comedo is an open, widely dilated follicle with black-colored sebum, due to melanin and oxidation, and keratinous material that forms a plug, thereby obstructing the pilosebaceous duct. A closed comedo is a closed follicle filled with impacted sebum covered by keratin that has a whitish color. A papule is a small, raised, red, dome-shaped palpable lesion. A pustule is a raised, dome-shaped palpable lesion containing yellow fluid (pus). A nodule may be a raised or deep-seated, dome-shaped palpable lesion of at least 5 millimeters in diameter.
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) Population: all randomized participants who received at least one application of investigational product. Only those participants with data available at the specified time point were analyzed. Analysis was based on an analysis of covariance (ANCOVA) model with terms for Baseline value, treatment, and center.
Measure: Least Squares Mean (Standard Error); unit: Lesion counts
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 177 | 182
Lesion counts | -42.9 (1.93) | -22.0 (1.89)
Statistical Analysis 1: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -21.0, 95% CI 2-sided [-26.2 to -15.8]

2. Secondary Outcome: Absolute Change in Total Lesion Counts From Baseline to Weeks 1, 2, 4, and 8
Description: The investigator/subinvestigator counted all inflammatory lesions (papules, pustules, and nodular lesions) and non-inflammatory lesions (open and closed comedo) on the face at each study visit. An open comedo is an open, widely dilated follicle with black-colored sebum, due to melanin and oxidation, and keratinous material that forms a plug, thereby obstructing the pilosebaceous duct. A closed comedo is a closed follicle filled with impacted sebum covered by keratin that has a whitish color. A papule is a small, raised, red, dome-shaped palpable lesion. A pustule is a raised, dome-shaped palpable lesion containing yellow fluid (pus). A nodule may be a raised or deep-seated, dome-shaped palpable lesion of at least 5 millimeters in diameter.Data were analyzed using an ANCOVA model with terms for Baseline value, treatment, and center.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Lesion counts
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 178 | 182
Lesion counts
  Week 1, n=175, 179 | -15.9 (1.38) | -8.3 (1.35)
  Week 2, n=177, 182 | -24.4 (1.60) | -13.3 (1.57)
  Week 4, n=177, 182 | -32.0 (1.68) | -16.8 (1.65)
  Week 8, n=177, 182 | -39.6 (1.79) | -20.1 (1.75)
Statistical Analysis 1: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 1
Statistical Analysis 2: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 2
Statistical Analysis 3: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 4
Statistical Analysis 4: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 8

3. Secondary Outcome: Absolute Change From Baseline in Inflammatory Lesion (IL) Count and Non-inflammatory Lesion (NIL) Count to Weeks 1, 2, 4, 8, and 12
Description: The investigator/subinvestigator counted all inflammatory lesions (papules, pustules, and nodular lesions) and non-inflammatory lesions (open and closed comedo) on the face at each study visit. An open comedo is an open, widely dilated follicle with black-colored sebum, due to melanin and oxidation, and keratinous material that forms a plug, thereby obstructing the pilosebaceous duct. A closed comedo is a closed follicle filled with impacted sebum covered by keratin that has a whitish color. A papule is a small, raised, red, dome-shaped palpable lesion. A pustule is a raised, dome-shaped palpable lesion containing yellow fluid (pus). A nodule may be a raised or deep-seated, dome-shaped palpable lesion of at least 5 millimeters in diameter. Data were analyzed using an ANCOVA model with terms for Baseline value, treatment, and center.
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Lesion counts
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 178 | 182
Lesion counts
  IL, Week 1, n=175, 179 | -8.2 (0.68) | -4.6 (0.67)
  IL, Week 2, n=177, 182 | -12.3 (0.81) | -5.8 (0.79)
  IL, Week 4, n=177, 182 | -14.9 (0.83) | -8.4 (0.82)
  IL, Week 8, n=177, 182 | -16.8 (0.90) | -7.8 (0.88)
  IL, Week 12, n=177, 182 | -18.3 (0.90) | -9.6 (0.88)
  NIL, Week 1, n=175, 179 | -7.7 (1.08) | -3.7 (1.06)
  NIL, Week 2, n=177, 182 | -12.2 (1.27) | -7.5 (1.25)
  NIL, Week 4, n=177, 182 | -17.1 (1.32) | -8.4 (1.30)
  NIL, Week 8, n=177, 182 | -22.8 (1.38) | -12.3 (1.35)
  NIL, Week 12, n=177, 182 | -24.6 (1.54) | -12.3 (1.51)
Statistical Analysis 1: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 1; IL
Statistical Analysis 2: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 2; IL
Statistical Analysis 3: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 4; IL
Statistical Analysis 4: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 8; IL
Statistical Analysis 5: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 12; IL
Statistical Analysis 6: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p = 0.007, ANCOVA — Week 1; NIL
Statistical Analysis 7: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p = 0.008, ANCOVA — Week 2; NIL
Statistical Analysis 8: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 4; NIL
Statistical Analysis 9: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 8; NIL
Statistical Analysis 10: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 12; NIL

4. Secondary Outcome: Percent Change From Baseline in Total, Inflammatory, and Non-inflammatory Lesion Counts to Weeks 1, 2, 4, 8, and 12
Description: The percent change from Baseline to Weeks 1, 2, 4, 8, and 12 in lesion counts (total [inflammatory and non-inflammatory], inflammatory [IL], and non-inflammatory [NIL]) was analyzed using an ANOVA model with terms for treatment and center. Percent change from Baseline was calculated as: (post-Baseline value minus Baseline value) * 100.
Time Frame: Baseline; Weeks 1, 2, 4 and 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change in lesion counts
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 178 | 182
Percent change in lesion counts
  Total, Week 1, n=175, 179 | -22.26 (1.705) | -12.07 (1.676)
  Total, Week 2, n=177, 182 | -36.17 (2.052) | -19.63 (2.014)
  Total, Week 4, n=177, 182 | -45.43 (2.177) | -24.50 (2.137)
  Total, Week 8, n=177, 182 | -55.40 (2.378) | -27.43 (2.334)
  Total, Week 12, n=177,182 | -59.79 (2.754) | -30.15 (2.704)
  IL, Week 1, n=175, 179 | -30.85 (2.379) | -16.78 (2.338)
  IL, Week 2, n=177, 182 | -46.40 (2.720) | -20.74 (2.670)
  IL, Week 4, n=177, 182 | -54.38 (2.696) | -30.54 (2.647)
  IL, Week 8, n=177, 182 | -60.33 (2.810) | -28.02 (2.759)
  IL, Week 12, n=177,182 | -64.68 (2.859) | -36.16 (2.807)
  NIL, Week 1, n=175, 179 | -16.99 (2.127) | -7.92 (2.091)
  NIL, Week 2, n=177, 182 | -29.78 (2.570) | -17.93 (2.523)
  NIL, Week 4, n=177, 182 | -39.88 (2.584) | -19.72 (2.536)
  NIL, Week 8, n=177, 182 | -51.64 (2.923) | -25.86 (2.869)
  NIL, Week 12, n=177,182 | -55.17 (3.533) | -26.36 (3.468)
Statistical Analysis 1: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 1; Total
Statistical Analysis 2: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 2; Total
Statistical Analysis 3: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 4; Total
Statistical Analysis 4: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 8; Total
Statistical Analysis 5: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 12; Total
Statistical Analysis 6: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 1; IL
Statistical Analysis 7: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 2; IL
Statistical Analysis 8: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 4; IL
Statistical Analysis 9: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 8; IL
Statistical Analysis 10: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 12; IL
Statistical Analysis 11: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p = 0.002, ANCOVA — Week 1; NIL
Statistical Analysis 12: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 2; NIL
Statistical Analysis 13: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 4; NIL
Statistical Analysis 14: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 8; NIL
Statistical Analysis 15: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 12; NIL

5. Secondary Outcome: Number of Participants Who Had a Minimum 2-grade Improvement in the Investigator's Static Global Assessment (ISGA) Score From Baseline to Week 12
Description: Investigators evaluated the acne severity of the participants' face using the ISGA scale, ranging from 0 to 5: 0=clear skin with no inflammatory lesions (ILs) or non-inflammatory lesions (NILs); 1=almost clear: rare NILs with no more than rare papules; 2=mild acne: greater than Grade 1, some NILs with no more than a few ILs (papules/pustules only, no nodular lesions [NLs]); 3=moderate acne: greater than Grade 2, up to many NILs and had some ILs, but no more than one small NL; 4=severe acne: greater than Grade 3, up to many NILs and ILs, but no more than a few NLs; 5=very severe acne: many NILs and ILs and more than a few NLs, had cystic lesions.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants with data available at the specified time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 164 | 166
Participants | 31 | 2
Statistical Analysis 1: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Number of Participants Who Had an ISGA Score of 0 or 1 at Weeks 1, 2, 4, 8, and 12
Description: as for outcome 5
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 178 | 182
Participants
  Week 1, n=175, 179 | 4 | 1
  Week 2, n=177, 179 | 6 | 0
  Week 4, n=176, 178 | 12 | 1
  Week 8, n= 168, 173 | 16 | 3
  Week 12, n=164, 166 | 35 | 3
Statistical Analysis 1: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p = 0.174, ANCOVA — Week 1
Statistical Analysis 2: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p = 0.013, ANCOVA — Week 2
Statistical Analysis 3: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p = 0.001, ANCOVA — Week 4
Statistical Analysis 4: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p = 0.001, ANCOVA — Week 8
Statistical Analysis 5: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 12

7. Secondary Outcome: Number of Participants Who Had a Reduction in Total Lesions of at Least 50% From Baseline to Weeks 1, 2, 4, 8, and 12
Description: The proportion of participants who have a reduction in total lesions (inflammatory and non-inflammatory) of at least 50% from Baseline at Weeks 1, 2, 4, 8, and 12 was measured.
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 178 | 182
Participants
  Week 1, n=175, 179 | 25 | 7
  Week 2, n=177, 182 | 60 | 32
  Week 4, n=177, 182 | 86 | 38
  Week 8, n= 177, 182 | 115 | 54
  Week 12, n=177, 182 | 116 | 73
Statistical Analysis 1: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 1
Statistical Analysis 2: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 2
Statistical Analysis 3: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 4
Statistical Analysis 4: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 8
Statistical Analysis 5: Comparison: GI148512 vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Week 12

8. Secondary Outcome: Mean Change From Baseline in Erythema, Dryness, and Peeling Scores at Weeks 1, 2, 4, 8, 12/Withdrawal
Description: Erythema (redness), dryness, and peeling were evaluated independently by the investigator as: 0 (absent)=no erythema, dryness, or peeling; 1 (slight)=faint red/pink coloration, barely perceptible dryness with no flakes or fissure, mild localized peeling; 2 (mild)=light red/pink coloration, perceptible dryness with no flakes/fissure, mild and diffuse peeling; 3 (moderate)=medium red coloration, easily noted dryness and flakes but no fissure, moderate and diffuse peeling; 4 (severe)=beet red coloration, dryness with flakes and fissure, prominent dense peeling. Change from Baseline was calculated as the post-Baseline/Withdrawal value minus the Baseline value.
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12 or Withdrawal
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points/for different parameters, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 178 | 182
Scores on a scale
  Erythema, Week 1, n=177, 181 | -0.03 (0.53) | -0.13 (0.53)
  Erythema, Week 2, n=177, 176 | -0.07 (0.62) | -0.19 (0.61)
  Erythema, Week 4, n=173, 174 | -0.13 (0.68) | -0.20 (0.66)
  Erythema, Week 8, n= 164, 168 | -0.19 (0.61) | -0.23 (0.70)
  Erythema, Week 12, n=164, 167 | -0.19 (0.74) | -0.26 (0.70)
  Erythema, Withdrawal, n=12, 15 | 1.17 (1.80) | 0.47 (0.99)
  Dryness, Week 1, n=177, 181 | 0.16 (0.62) | -0.08 (0.36)
  Dryness, Week 2, n=177, 176 | 0.14 (0.56) | -0.06 (0.38)
  Dryness, Week 4, n=173, 174 | 0.06 (0.52) | -0.06 (0.39)
  Dryness, Week 8, n=164, 168 | 0.00 (0.46) | -0.08 (0.46)
  Dryness, Week 12, n=164, 167 | -0.04 (0.53) | -0.11 (0.44)
  Dryness, Withdrawal, n=12, 15 | 0.58 (1.24) | 0.33 (1.11)
  Peeling, Week 1, n=177, 181 | 0.01 (0.43) | -0.03 (0.29)
  Peeling, Week 2, n=177, 176 | 0.02 (0.50) | -0.03 (0.31)
  Peeling, Week 4, n=173, 174 | -0.01 (0.41) | 0.00 (0.32)
  Peeling, Week 8, n=164, 168 | -0.01 (0.48) | -0.01 (0.35)
  Peeling, Week 12, n=164, 167 | -0.02 (0.51) | -0.05 (0.27)
  Peeling, Withdrawal, n=12, 15 | 0.42 (0.90) | 0.13 (0.92)

9. Secondary Outcome: Mean Change From Baseline in Itching and Burning/Stinging Scores at Weeks 1, 2, 4, 8, 12/Withdrawal
Description: Itching and burning/stinging were evaluated by the participant as: 0 (none)=normal, no discomfort; 1 (slight)=noticeable discomfort that caused intermittent awareness; 2 (mild)=noticeable discomfort that caused continuous awareness; 3 (moderate)=noticeable discomfort that caused intermittent awareness and interfered occasionally with normal daily activities; 4 (severe)=definite continuous discomfort that interfered with normal daily activities. Change from Baseline was calculated as the post-Baseline/Withdrawal value minus the Baseline value.
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12 or withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GI148512 | Vehicle Gel
Number analyzed (Participants) | 178 | 182
Scores on a scale
  Itching, Week 1, n=177, 181 | -0.01 (0.45) | -0.12 (0.48)
  Itching, Week 2, n=177, 176 | 0.01 (0.48) | -0.13 (0.53)
  Itching, Week 4, n=173, 174 | 0.01 (0.60) | -0.14 (0.54)
  Itching, Week 8, n=164, 168 | -0.04 (0.51) | -0.11 (0.52)
  Itching, Week 12, n=164, 167 | -0.07 (0.44) | -0.12 (0.52)
  Itching, Withdrawal, n=12, 15 | 1.33 (1.44) | 0.20 (1.21)
  Burning/Stinging, Week 1, n=177, 181 | 0.15 (0.49) | -0.04 (0.29)
  Burning/Stinging, Week 2, n=177, 176 | 0.15 (0.58) | -0.03 (0.34)
  Burning/Stinging, Week 4, n=173, 174 | 0.05 (0.42) | -0.02 (0.40)
  Burning/Stinging, Week 8, n=164, 168 | 0.04 (0.37) | -0.02 (0.44)
  Burning/Stinging, Week 12, n=164, 167 | 0.05 (0.49) | -0.04 (0.38)
  Burning/Stinging,Withdrawal, n=12, 15 | 1.00 (1.21) | 0.73 (1.39)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs collected from the start of study treatment until Week 12 or premature withdrawal are reported.
Description: SAEs and non-serious AEs are reported for members of the ITT Population,comprised of all randomized participants who received at least one application of investigational product.
Arm/Group | GI148512 | Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 0/178 | 0/182
Other Adverse Events (participants affected / at risk) | 78/178 | 61/182
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GI148512 (N=178) | Vehicle Gel (N=182)
Nasopharyngitis (Infections and infestations) | 40 | 53
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 16 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 4
Erythema (Skin and subcutaneous tissue disorders) | 10 | 2
Facial pain (General disorders) | 19 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.